CLINICAL TRIAL: NCT00000855
Title: The Safety, Tolerance, and Pharmacokinetics of Zidovudine in Premature Infants Exposed to HIV.
Brief Title: A Study to Evaluate the Safety and Tolerability of Zidovudine (ZDV) in Premature Infants Born to HIV-Positive Women.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 331; 11303 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Zidovudine; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
The purpose of this study is to examine the safety and tolerability of ZDV when given to premature infants born to HIV-positive women to prevent HIV infection.

ZDV has been used successfully to prevent the transmission of HIV from mother to child during pregnancy and birth. However, ZDV has been given to very few premature babies, and the best dose to use has not yet been determined.

DETAILED DESCRIPTION:
In the preliminary group of premature infants, those receiving q 6h dosing had an average trough concentration of 7.3 uM (18%). However, the premature infants in the preliminary pharmacokinetic study did not have long term follow-up to assess toxicity. Due to the potential for altered ZDV pharmacokinetics and increased toxicity in this population, an evaluation of ZDV pharmacokinetics in premature infants is proposed.

Premature infants less than or equal to 34 weeks gestational age at birth and begun on ZDV by their clinical caregivers will be entered into the protocol within the first 5 days of life. Upon entry, ZDV will be administered every 12 hours intravenously or orally. The study will require 9 serum samples for ZDV assay collected over 30 days, some additional clinical laboratory tests collected over 12 weeks, collection of 3 spot urine samples, and collection of routine clinical data.

ELIGIBILITY:
Inclusion Criteria

Your baby may be eligible for this study if he/she:

* Requires ZDV (as decided by your doctor) because you are HIV-positive.
* Is 1-5 days old and was born prematurely.

Exclusion Criteria

Your baby will not be eligible for this study if he/she:

* Is not expected to live 6 weeks because of severe illness.
* Is having problems with blood pressure or is not urinating enough.

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35
Dates: Study Completion 2000-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirochnick M, Study Chair; Dankner D, Study Chair; Capparelli E, Study Chair
Locations (36):
- United States (35):
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Phoenix Childrens Hosp, Phoenix, Arizona
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Univ of Florida Gainesville, Gainesville, Florida
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Univ of Chicago Children's Hosp, Chicago, Illinois
  - Division of Inf Diseases/ Indiana Univ Hosp, Indianapolis, Indiana
  - Children's Hosp of Boston, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - Univ of Rochester Med Ctr, Rochester, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Westchester Hosp, Valhalla, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Med Univ of South Carolina, Charleston, South Carolina
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Children's Hosp of the King's Daughters, Norfolk, Virginia
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan, Puerto Rico

REFERENCES:
- [Background] Capparelli EV, Mirochnick M, Dankner WM, Blanchard S, Mofenson L, McSherry GD, Gay H, Ciupak G, Smith B, Connor JD; Pediatric AIDS Clinical Trials Group 331 Investigators. Pharmacokinetics and tolerance of zidovudine in preterm infants. J Pediatr. 2003 Jan;142(1):47-52. doi: 10.1067/mpd.2003.mpd0335. PMID 12520254